CLINICAL TRIAL: NCT00146848
Title: Pacing Evaluation - Atrial Support Study in Cardiac Resynchronization Therapy
Brief Title: PEGASUS CRT Study: Atrial Support Study in Cardiac Resynchronization Therapy
Acronym: PEGASUS CRT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-CA-100604-H; PEGASUS
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Results first posted 2010-09-23 (Estimated); Last update posted 2011-12-28 (Estimated); Status verified 2011-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DDD-40 (Active Comparator): DDD-40 for this trial is the comparator arm. Even though patients are receiving a CRT-D device, atrial support pacing in this arm will be limited as the device will not pace unless the rate falls below 40 bpm.
  Interventions: Device: Atrial support pacing through cardiac resynchronization therapy. Device: RENEWAL family of CRT-D devices
- DDDR-40 (Active Comparator): DDDR-40 programming will initiate atrial support pacing if the rate falls below 40 bpm or if atrial support is needed in response to increased activity.
  Interventions: Device: Atrial support pacing through cardiac resynchronization therapy. Device: RENEWAL family of CRT-D devices
- DDD-70 (Active Comparator): Atrial support pacing in this arm will be delivered when the rate falls below 70 bpm.
  Interventions: Device: Atrial support pacing through cardiac resynchronization therapy. Device: RENEWAL family of CRT-D devices

INTERVENTIONS:
Device: Atrial support pacing through cardiac resynchronization therapy. Device: RENEWAL family of CRT-D devices — All subjects in this trial receive the same device. For the purpose of this trial, "intervention" is programming mode and lower rate limit to deliver atrial support pacing in the two treatment arms, while the control arm will receive programming where limited atrial support pacing is delivered. DDD-70 and DDDR-40 are the treatment arms programmed to receive atrial support pacing and will be compared to the DDD-40 arm.

SUMMARY:
This study will look at different pacing modes (how a device is programmed to pace one's heart), and how these modes may assist in one's daily activities and how one is feeling.

DETAILED DESCRIPTION:
PEGASUS CRT is a multicenter trial that will assess the effect of a cardiac resynchronization therapy defibrillator (CRT-D) device programmed to DDD-70 or DDDR-40 compared to a CRT device programmed to DDD-40 in heart failure patients. The effect of atrial support pacing in heart failure patients will be assessed using a clinical composite rating. A sub-study will evaluate the effect pacing mode has on exercise capacity in this heart failure population.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet current indications for the CONTAK RENEWAL® family of cardiac resynchronization therapy defibrillator (CRT-D) devices or future Food and Drug Administration (FDA) approved Guidant CRT-D devices
* Patients who sign and date a Patient Informed Consent at, or prior to, the implant visit
* Patients who are in sinus rhythm at the time of implant
* Patients who remain in the clinical care of the enrolling physician in approved centers
* Patients who are on optimal pharmacologic therapy or who have developed a recent implantable cardioverter defibrillator (ICD) indication that necessitates ICD therapy concurrent with the optimization of pharmacologic therapy

Exclusion Criteria:

* Patients whose medical condition is expected to preclude the use of the protocol-required pacing mode (dual chamber pacing [DDD or DDDR]) and respective lower rate limits
* Patients with permanent atrial fibrillation or atrial flutter
* Patients who are in complete heart block
* Patients who have previously had a pacemaker, ICD, or CRT device
* Patients whose life expectancy is less than 12 months due to other medical conditions
* Patients who are expected to receive a heart transplant during the duration of the study
* Patients who have other cardiac surgeries or procedures planned but not yet performed
* Patients who currently have or who are likely to receive a tricuspid valve prosthesis
* Patients who are currently enrolled in another investigational study or registry that would directly impact the treatment or outcome of the current study.
* Patients who are younger than 18 years of age
* Patients who are mentally incompetent and cannot sign a Patient Informed Consent form or comply with the study
* Patients who are or become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1742 (Actual)
Dates: Start 2004-12; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David O. Martin, MD, MPH, Principal Investigator — The Cleveland Clinic; John Day, Principal Investigator — Utah Heart Clinic, LDS Hospital
Locations (1):
- The Cleveland Clinic Hospital, Cleveland, Ohio, United States

REFERENCES:
- [Background] Martin DO, Stolen KQ, Brown S, Yu Y, Christie C, Doshi SK, Smith JM, Gold MR, Day JD. Pacing Evaluation-Atrial SUpport Study in Cardiac Resynchronization Therapy (PEGASUS CRT): design and rationale. Am Heart J. 2007 Jan;153(1):7-13. doi: 10.1016/j.ahj.2006.10.013. PMID 17174627
- [Derived] Martin DO, Day JD, Lai PY, Murphy AL, Nayak HM, Villareal RP, Weiner S, Kraus SM, Stolen KQ, Gold MR. Atrial support pacing in heart failure: results from the multicenter PEGASUS CRT trial. J Cardiovasc Electrophysiol. 2012 Dec;23(12):1317-25. doi: 10.1111/j.1540-8167.2012.02402.x. Epub 2012 Jul 25. PMID 22830441

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began on November 8, 2004, was completed on December 21, 2007, with study follow-up commencing January 30, 2009. This trial was conducted at institutional settings throughout the United States and Australia.
Pre-assignment Details: All patients with successful system implants were programmed to DDD-40 (atrial rate support above 40 bpm; limited atrial pacing) for the first 6-weeks of the trial. Randomization (1:1:1 allocation) occurred after patients had reached the 6-week visit and continued to meet all of the eligibility criteria for the trial.
Groups:
- DDD-40: Atrial Tracking (atrial rate support above 40 bpm)
- DDD-70: Atrial Rate Support (atrial rate support above 70 bpm)
- DDDR-40: Rate Adaptive Pacing (atrial rate support above 40 bpm with rate responsive pacing)
Period: Pre-randomization
Arm/Group | DDD-40 | DDD-70 | DDDR-40
Started | 1742 (Registered) | 0 | 0
Completed | 1433 (Reached 6-week visit and were randomized) | 0 | 0
Not Completed | 309 | 0 | 0
Not completed — Death | 19 | 0 | 0
Not completed — Lost to Follow-up | 70 | 0 | 0
Not completed — Physician Decision | 8 | 0 | 0
Not completed — Protocol Violation | 172 | 0 | 0
Not completed — Withdrawal by Subject | 40 | 0 | 0
Period: Post-randomization
Arm/Group | DDD-40 | DDD-70 | DDDR-40
Started | 475 | 488 | 470
Completed | 437 | 441 | 431
Not Completed | 38 | 47 | 39
Not completed — Lost to Follow-up | 12 | 15 | 12
Not completed — Withdrawn | 26 | 32 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DDD-40 | DDD-70 | DDDR-40 | Total
Number analyzed (Participants) | 475 | 488 | 470 | 1433
Age Continuous [Mean (Standard Deviation); unit: years] | 67.3 (11.4) | 67.5 (10.4) | 66.7 (11.6) | 67.2 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165 | 156 | 165 | 486
  Male | 310 | 332 | 305 | 947

OUTCOME MEASURES:

1. Secondary Outcome: Change in Quality of Life
Description: Quality of Life as assessed by the Minnesota Living with Heart Failure Questionniare for those patients with paired data at 6 weeks and 12 months. This score is on a scale of 0(best)- 105(worst). A negative change denotes improvement.
Time Frame: From randomization (6-weeks) through 12-month visit
Population: Quality of Life was analyzed for those patients with paired data available at the 6 week and 12 month visit. Patients were analyzed in their randomized groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DDD-40 | DDD-70 | DDDR-40
Number analyzed (Participants) | 348 | 370 | 357
units on a scale | -2.97 (24.18) | -3.27 (22.77) | -4.46 (25.43)
Statistical Analysis 1: Comparison: DDD-40 vs DDD-70; The changes in quality of life were compared between groups using two-sided t-tests; Test type: Superiority or Other; p = 0.86, t-test, 2 sided; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [-3.14 to 3.74], Standard Error of Mean 1.75
Statistical Analysis 2: Comparison: DDD-40 vs DDDR-40; The difference in changes in quality of life between groups were compared using a t-test; Test type: Superiority or Other; p = 0.43, t-test, 2 sided; Mean Difference (Final Values) = 1.49, 95% CI 2-sided [-2.18 to 5.16], Standard Error of Mean 1.87

2. Primary Outcome: Clinical Composite Score
Description: The primary outcome measure classified patients as improved, unchanged or worsened, based on a 4 components clinical composite score using the following four components: death, heart failure hospitalization, New York Heart Association [NYHA] class, patient's Global Assessment rating. Best value is improved, whereas worst value is worsened.
Time Frame: From randomization (6-weeks) through 12-month visit
Population: This analysis is intention to treat (ITT) in terms of patient's being analyzed according to their randomized group. Last observation carried forward (LOCF) method was used for missing NYHA and global assessment measures at 12 months.
Measure: Number; unit: participants
Arm/Group | DDD-40 | DDD-70 | DDDR-40
Number analyzed (Participants) | 437 | 441 | 431
participants
  Improved | 230 | 235 | 229
  Unchanged | 84 | 94 | 85
  Worsened | 123 | 112 | 117
Statistical Analysis 1: Comparison: DDD-40 vs DDD-70; One sided test testing for shift towards improvement in either atrial support pacing treatment arm compared to the DDD-40 arm; Test type: Superiority or Other; p = 0.55, Cochran-Armitage test for trend
Statistical Analysis 2: Comparison: DDD-40 vs DDDR-40; Test type: Superiority or Other; p = 0.80, Cochran-Armitage test for trend

3. Secondary Outcome: Change in Self Assessed Physical Activity
Description: Physical activity was assessed using the Physical Activity Scale of the Elderly (PASE) questionnaire for those patients with paired data available at the 6 week and 12 month visits. The PASE is designed to assess physical activity in older persons. The total PASE score was computed by multiplying the amount of time spent in each activity (hours/week) or participation (yes/no) in an activity by empirically derived item weights and summing over all activities. PASE scores for this study ranged from 0 to 756 with higher scores indicating more physical activity.
Time Frame: From randomization (6-weeks) through 12-month visit
Population: Physical activity was assessed using the Physical Activity Scale for the Elderly and was analyzed for those patients with paired data available at the 6 week and 12 month visit. Patients were analyzed in their randomized groups. Postive values for changes denote improvements.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DDD-40 | DDD-70 | DDDR-40
Number analyzed (Participants) | 339 | 362 | 348
units on a scale | 12.45 (78.62) | 22.62 (88.86) | 25.69 (92.41)
Statistical Analysis 1: Comparison: DDD-40 vs DDD-70; Compare the difference in the changes in physical activity scores between groups using a t-test; Test type: Superiority or Other; p = 0.11, t-test, 2 sided; Mean Difference (Final Values) = -10.17, 95% CI 2-sided [-22.65 to 2.30], Standard Error of Mean 6.35
Statistical Analysis 2: Comparison: DDD-40 vs DDDR-40; Compare the difference in the changes in physical activity scores between groups using a t-test. To adjust for multiple comparisons, an alpha level of 0.025 should be used to deem significance; Test type: Superiority or Other; p = 0.04, t-test, 2 sided; Mean Difference (Final Values) = -13.24, 95% CI 2-sided [-26.11 to -0.37], Standard Error of Mean 6.55

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from randomization (6-weeks) through the 12-month follow-up visit. Per trial design, serious adverse events were not collected in this trial.
Description: Source vocabulary for AE coding was not used in this trial. Serious adverse events were not collected in this trial per trial design.
Arm/Group | DDD-40 | DDD-70 | DDDR-40
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 129/475 | 119/488 | 112/470
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DDD-40 (N=475) | DDD-70 (N=488) | DDDR-40 (N=470)
Cardiovascular related (Cardiac disorders) | 80 (124) | 89 (125) | 76 (117)
Non-device, non-lead, non-procedure or non-cardiovascular related AE "other" (General disorders) | 64 (82) | 43 (58) | 45 (54)

LIMITATIONS AND CAVEATS:
Lack of longer-term follow-up. Single blind design where investigator could be aware of treatment assignment. Two conservative atrial support pacing modes; results should not be extended to substantially more atrial pacing and higher heart rates.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 30 days from the time submitted to the sponsor for review.